CLINICAL TRIAL: NCT04049331
Title: Improving Patient-Important Outcomes With Testosterone Replacement in Hypogonadal Men With a Prior History of Cancer
Brief Title: Testosterone Replacement in Male Cancer Survivors With Fatigue and Low Testosterone
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01751
Record Dates: First submitted 2019-07-23; First posted 2019-08-08 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Hypogonadism, Male; Fatigue Syndrome, Chronic
Keywords: testosterone; hypogonadism; cancer related fatigue
MeSH Terms: conditions — Eunuchism; Fatigue Syndrome, Chronic; Hypogonadism | interventions — testosterone undecanoate; Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Testosterone (Experimental): Testosterone undecanoate injection 750 MG/3 ML
  Interventions: Drug: Testosterone Undecanoate 750 MG/3 ML Intramuscular Solution [AVEED]
- Placebo (Placebo Comparator): clinical grade saline 0.9% sodium chloride injection
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Testosterone Undecanoate 750 MG/3 ML Intramuscular Solution [AVEED] — first two doses four weeks apart; following three more doses every ten weeks.
  Other Names: study drug
  Arms: Testosterone
Other: placebo — first two doses four weeks apart; following three more doses every ten weeks.
  Arms: Placebo

SUMMARY:
The overall goal of this study is to evaluate the effect of a testosterone drug called Depo-Testosterone (or 'testosterone cypionate'), an FDA-approved drug for improving fatigue, sexual function, quality of life, body composition, muscle strength, and physical activity in young cancer survivors who report fatigue and have low testosterone. Main hypothesis is that Testosterone administration in young male cancer survivors who are in remission for at least 1 year, report cancer-related fatigue and have symptomatic testosterone deficiency will be associated with greater improvements in fatigue scores compared with placebo.

DETAILED DESCRIPTION:
The overall goal of this proposal is to evaluate the efficacy of testosterone replacement therapy in improving fatigue and other outcomes such as sexual function, quality of life, body composition, muscle strength and physical activity in a double-blind, randomized, placebo-controlled trial in young cancer survivors who report fatigue and have testosterone deficiency.

Fatigue is one of the most prevalent and debilitating symptoms in men with cancer affecting 70-100% of patients irrespective of their age. Cancer-related fatigue is experienced by patients not only during active cancer treatment, but is also highly prevalent in cancer survivors who exhibit persistent fatigue months to years after the end of their treatment with the highest prevalence being in recipients of chemotherapy and/or radiation therapy.

In addition to fatigue, sexual dysfunction is also highly prevalent in male cancer survivors. Male cancer survivors also have increased fat mass and decreased lean body mass, a phenotype that predisposes them to reduced muscle strength. This phenotype of fatigue, sexual dysfunction and adverse body composition is commonly encountered in non-cancer patient populations with testosterone deficiency, a condition which is also highly prevalent (50-90%) in cancer survivors. Pivotal trials of testosterone replacement therapy in non-cancer patient populations have shown an improvement in fatigue, sexual function and body composition in men randomized to testosterone compared with placebo. However, the efficacy of testosterone replacement therapy on cancer-related fatigue has not been studied.

ELIGIBILITY:
Inclusion Criteria:

* Cancer survivors who have received chemotherapy and/or radiation therapy for their cancer and are now in remission for at least one year
* Non-hormone-dependent cancer, including most solid tumors, lymphomas and leukemias
* Age: 18-54 years
* Serum testosterone, measured by mass spectrometry (gold standard method), of <348 ng/dl and/or free testosterone <70 pg/ml. The lower limits of the normal range for total testosterone in healthy young men (age 19-40 years), is 348 ng/dL and the lower limits of free testosterone is <70 pg/ml in the Framingham Heart Study sample97. Therefore, young symptomatic men with total testosterone <348 ng/dl could be considered testosterone deficient. As sex hormone binding globulin levels may be elevated in some men with cancer (resulting in elevation in total testosterone level), some of these symptomatic men may still be hypogonadal despite having total testosterone above this cut-off limit. However; their free testosterone levels may still be below the lower limit of normal. Thus, we will also include men with free testosterone <70 pg/mL.
* Self-reported fatigue. We have selected these symptoms because they are commonly reported in male cancer survivors. Fatigue will be defined as a score on Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) subscale of <40, which best divides cancer patients from the general population with 84% accuracy, and was used as the cut-off for the NIA-funded 50-million-dollar testosterone trial (The T-Trial).
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Men with hormone-dependent cancers (breast, prostate or adenocarcinoma of unknown origin)
* Men with brain cancer (potential cognitive impairment)
* Use of anabolic agents (testosterone, dehydroepiandrosterone, growth hormone) within the past 6 months
* Appetite stimulating agents e.g. megestrol acetate within the past 6 months
* Systemic glucocorticoids e.g. prednisone 20 mg daily or equivalent doses of other glucocorticoids for more than two weeks in the past 6 months
* Baseline hematocrit >48%
* PSA >4 ng/ml in Caucasians; >3 ng/ml in African-Americans
* Men with 1st order relatives with a history of prostate cancer
* Uncontrolled congestive heart failure
* Severe untreated sleep apnea
* Myocardial infarction, acute coronary syndrome, revascularization surgery, or stroke within 3 months

  o Previous stroke with residual cognitive or functional deficits; Mini-Mental State Examination score <24
* Serum creatinine >2.5 mg/dL; ALT 3x upper limit of normal
* Poorly controlled diabetes as defined by hemoglobin A1c >8.5%; Body mass index (BMI) >45 kg/m2
* Untreated unipolar depression (treated depression with medications or counseling will be allowed
* Bipolar disorder or schizophrenia

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-03-22 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Fatigue change | 9 months
  (Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F) questionnaire

SECONDARY OUTCOMES:
Sexual function change | 9 months
  Harbor-UCLA 7-day Sexual Function Questionnaire
Sexual function change | 9 months
  International Index of Erective Function (IIEF) questionnaire
Body composition change | 9 months
  Lean body mass and fat mass (kg) measured by dual energy x-ray absorptiometry (DEXA)
Changes to mood and well-being | 9 months
  Mood and well-being will be assessed by the Positive and Negative Affect Scale (PANAS) affectivity balance scale, which includes 10 questions each for Positive Affect and Negative Affect. Many behavioral scientists consider affectivity as the cleanest window on an individual's wellbeing. The most sensitive indicator of impaired wellbeing has been shown to be affective dysregulation, which is reflected in affectivity balance. The latter incorporates negative affects (e.g., anxiety, depression) as well as positive affects (e.g., joy).
Muscle strength change | 9 months
  Maximal voluntary muscle strength in the lower extremities will be assessed by conducting the leg press exercise by the 1-repetition maximum method and assessing loaded stair climb power.
Sleep quality change | 9 months
  Pittsburgh Sleep Quality Index (PSQI)
Sleep quality change | 9 months
  Insomnia Severity Index (ISI)
Sleep quality change | 9 months
  Actigraphy
Daily physical activity change | 9 months
  Validated triaxial accelerometry (actigraphy)

CONTACTS AND LOCATIONS:
Overall Officials: Jose M Garcia, MD, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Veterans Affairs Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No